CLINICAL TRIAL: NCT03372460
Title: Combined Transcranial Direct Current Stimulation and Virtual Reality for PTSD
Brief Title: tDCS Plus Virtual Reality for PTSD
Acronym: TAVRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: D2450-R; 2017-053 (Other: PVAMC IRB); 1633742 (Other: PVAMC IRB)
Record Dates: First submitted 2017-11-03; First posted 2017-12-13 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Post-Traumatic Stress Disorder
Keywords: Transcranial Direct Current Stimulation; Stress Disorders, Post-Traumatic; Virtual Reality; Prefrontal Cortex; Veterans; Quality of Life
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants are assigned to receive either active or sham stimulation during the tDCS+VR sessions in parallel for the duration of the study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blind tDCS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active Stimulation (Active Comparator): Active stimulation (tDCS) will be used in the dose of 2mA /25 min per day, for 6 sessions over the course of 2 weeks (3 sessions per week).
  Interventions: Device: Active stimulation; Other: Virtual Reality (VR)
- Sham Stimulation (Sham Comparator): Sham tDCS uses the device study mode (10 µA over 15 ms current pulse applied every 550 ms, 3ms peak current). This process will be used for each of the 6 sessions during a 2 week period.
  Interventions: Device: Sham stimulation; Other: Virtual Reality (VR)

INTERVENTIONS:
Device: Active stimulation — For active tDCS, the investigators will use a 1x1 configuration with the anode placed over EEG coordinates AF7/Fp1/AF3 (using the 10-20 EEG convention) and the cathode between EEG coordinate OZ and the contralateral mastoid (covering approximately PO8/P8). The investigators will use 3x3 cm sponge covered electrodes and a 2mA current for 25 minutes per session.
  Other Names: Active tDCS
  Arms: Active Stimulation
Device: Sham stimulation — For sham tDCS, the investigators will use the same electrode and sponge configuration as active tDCS, but using the device study mode (10 µA over 15 ms current pulse applied every 550 ms, 3ms peak current).
  Other Names: Sham tDCS
  Arms: Sham Stimulation
Other: Virtual Reality (VR) — Participants will undergo VR exposure to trauma-related context.

SUMMARY:
This study tests the efficacy of combining non-invasive brain stimulation, called transcranial direct current stimulation (tDCS), with virtual reality exposure as a treatment for Veterans with chronic posttraumatic stress disorder (PTSD). Investigators tested whether this intervention improves PTSD symptoms and improves quality of life. Results from this study may be used to develop a new non-medication approach to treating chronic PTSD.

DETAILED DESCRIPTION:
PTSD is highly prevalent in Veterans and is associated with significant psychiatric and medical comorbidity, as well as poor quality of life. Despite its prevalence and impact, the success of currently available treatments is mixed, highlighting the need for novel approaches that aim to reduce symptoms and improve outcomes. Prior research demonstrated that reduced activity in a part of the brain, the ventromedial prefrontal cortex (VMPFC), is associated with an inability to regulate fear responses, preventing the generation of safety memories and allowing PTSD symptoms to persist. Targeting the VMPFC with non-invasive electrical brain stimulation may therefore alleviate these symptoms.

Transcranial direct current stimulation (tDCS) is a type of non-invasive brain stimulation that may enhance the likelihood of neuronal activity in the VMPFC. In doing so, tDCS prepares the brain to respond to external stimuli and to facilitate learning and memory. Because therapeutic success from exposure to trauma-related content - as used in exposure-based therapy for PTSD - is thought to be based on an adaptive learning process, applying tDCS in combination with exposure to trauma cues may effectively boost exposure-based learning. In this study, investigators at the VA Providence Healthcare System will use a standardized virtual reality (VR) setting to deliver trauma-related content. The virtual reality setting involves three, 8-minute driving scenarios, constituting one VR session, which consist of VR stimuli (sights, sounds, smells, etc.) often encountered in combat training and in theater.

Eligible participants will be randomized to receive six sessions of either active tDCS plus virtual reality (tDCS+VR) or sham tDCS+VR. Clinical and self-report assessments will be completed at baseline, midpoint, and endpoint, as well as 1 and 3 months following the final VR session. Primary outcome measures occur at the 1 month timepoint. Psychophysiology (skin conductance reactivity) will be collected throughout each VR session to capture habituation. Participants will also undergo a MRI before and after completion of all six active or sham tDCS+VR sessions to assess change over time. Additionally, MRI data will be used for electrical field modeling to predict treatment response based on individually obtained electrical field values in PTSD relevant neural circuitry. Participants may also choose to participate in an optional pre-active or sham tDCS+VR session EEG and an optional 1-month follow-up MRI.

ELIGIBILITY:
Inclusion Criteria:

* Must be a Veteran
* Located in the greater Providence and Boston areas
* Have a diagnosis of chronic PTSD, meeting DSM-5 criteria
* If in treatment, symptomatic despite ongoing stable treatment regimens for at least 6 weeks prior to study procedures.
* Willing and able to comply with all study related procedures and visits
* Capable of independently reading and understanding study materials and providing informed consent.

Exclusion Criteria:

Contraindications to MRI or tDCS, including:

* Implanted device (e.g., deep brain stimulation) or metal in the brain, cervical spinal cord, or upper thoracic spinal cord.
* Skin lesions at the site of stimulation that may increase conductance (e.g., vascular moles or angiomas)
* Pregnancy/lactation, or planning to become pregnant during the study
* Lifetime history of moderate or severe traumatic brain injury (TBI)
* Current unstable medical conditions
* Current (or past if appropriate) significant neurological disorder, or lifetime history of a) seizure disorder b) primary or secondary CNS tumors c) stroke or d) cerebral aneurysm.

Other exclusions:

* Primary psychotic disorder
* Bipolar I disorder
* Active moderate/severe substance use disorders (within the last month, excluding nicotine/caffeine)
* Active suicidal intent or plan as detected on screening instruments or in the investigative team's judgment is likely to attempt suicide within 6 months
* Other conditions or circumstances that, in the opinion of the investigator team, have the potential to prevent completion and/or have a confounding effect on outcome assessments.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2018-04-02 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noah S. Philip, MD, Principal Investigator — Providence VA Medical Center, Providence, RI
Locations (1):
- Providence VA Medical Center, Providence, RI, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van 't Wout-Frank M, Arulpragasam AR, Faucher C, Aiken E, Shea MT, Jones RN, Greenberg BD, Philip NS. Virtual Reality and Transcranial Direct Current Stimulation for Posttraumatic Stress Disorder: A Randomized Clinical Trial. JAMA Psychiatry. 2024 May 1;81(5):437-446. doi: 10.1001/jamapsychiatry.2023.5661. PMID 38446471

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Following enrollment, 10 Veterans were not randomized. Of these 10 Veterans, five were ineligible, three were lost to contact, and 2 were discontinued due to other concerns.
Period: Overall Study
Arm/Group | Active Stimulation | Sham Stimulation
Started | 26 | 29
Included in ITT Sample | 26 | 28 (1 Veteran discontinued due to stimulation site discomfort, not included in ITT sample.)
Completed All 6 VR Sessions | 21 (Two completed 3 VR sessions (1 family emergency but continued study, 1 had worsening symptoms and withdrew after assessments). Two completed 2 VR sessions (1 had site discomfort and withdrew after assessments, 1 was lost to contact). One completed 1 VR session, withdrew due to COVID-19 infection.) | 25 (One completed 5 VR sessions (change in health status but continued study), two completed four VR sessions (1 lost to contact, 1 had worsening symptoms and withdrew after assessments).)
Completed End-of-treatment Assessments | 24 | 27
Completed 1-month Follow-up | 19 (Five did not complete 1-month follow up. Of these, three were lost to contact and two were discontinued after completion of end-of-treatment assessments.) | 27
Completed 3-month Follow-up | 10 (Nine did not complete 3-month follow up. Of these, 4 were discontinued due to worsening symptoms or decision to pursue other treatment. Two were withdrawn by PI (1 no longer eligible, 1 unrelated SAE). Three were lost to contact.) | 19 (Eight did not complete 3-month follow-up. Of these, five were discontinued due to worsening symptoms or decision to pursue other treatment. Two were withdrawn by PI (1 due to increase in suicidal ideation, 1 unrelated SAE). One was lost to contact.)
Completed (Included in primary intent-to-treat (ITT) analysis (imputed)) | 26 | 28
Not Completed | 0 | 1
Not completed — Discontinued due to stimulation site discomfort | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Stimulation | Sham Stimulation | Total
Number analyzed (Participants) | 26 | 28 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 44 (12) | 47 (9) | 46 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 25 | 26 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 21 | 25 | 46
  Unknown or Not Reported | 3 | 0 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 21 | 22 | 43
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 26 | 28 | 54
PTSD Checklist for DSM-5 (PCL-5) [Mean (Standard Deviation); unit: score on a scale] — Total symptom severity score (range: 0-80) with higher scores indicating more severe PTSD symptoms.
  score on a scale | 48.6 (12.1) | 45.0 (11.9) | 46.72 (12.02)
Clinician-Administered PTSD Scale for DSM-5 [Mean (Standard Deviation); unit: score on a scale] — Total scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
  score on a scale | 44.8 (8.2) | 40.5 (8.1) | 42.59 (8.37)
Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ) [Mean (Standard Deviation); unit: score on a scale] — The 16-item QLESQ (short form) evaluates quality of life and other areas of change related to functioning outside of symptom domains (e.g., physical health, mood, leisure time activities, social relationships, etc.). Items are rated on how satisfied the respondent has been in the past week (1 = "very poor" to 5 = "very good "). A total raw score (range: 16-80). Higher outcomes indicate better quality of life, greater enjoyment, and satisfaction.
  score on a scale | 35.9 (8.9) | 39.2 (9.8) | 37.61 (9.42)
Social and Occupational Function Scale (SOFAS) [Mean (Standard Deviation); unit: score on a scale] — Scores range from 0 to 100, with higher scores indicating better social and occupational functioning.
  score on a scale | 40.5 (9.7) | 43.0 (11.2) | 42.20 (10.31)
Inventory of Depressive Symptomatology Self Report (IDSSR) [Mean (Standard Deviation); unit: score on a scale] — Total minimum score of 0 and a maximum score of 84. A higher score on the IDSSR indicates increased depressive symptom severity.
  score on a scale | 41.6 (12.0) | 38.6 (13.0) | 40.04 (12.52)

OUTCOME MEASURES:

1. Primary Outcome: Post-traumatic Stress Disorder Checklist for DSM-5 (PCL-5) Total Score
Description: The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. Items are rated on how much the symptom bothered the respondent in the past month (0 = "not at all bothered by" to 4 = "extremely bothered "). A total symptom severity score (range: 0-80) can be obtained by summing the scores for each of the 20 items, with higher scores indicating more severe PTSD symptoms. PCL-5 scores at 1 month was the primary symptom outcome measure for this study.
Time Frame: Baseline, Midpoint (1 week after VR session 3), Endpoint (2 weeks after VR session 6), 1 Month Follow-up, 3 Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 48.6 (12.1) | 45.0 (11.9)
  Midpoint | 38.5 (14.4) | 41.3 (15.1)
  Endpoint | 36.0 (15.4) | 38.9 (15.1)
  1 Month Follow-Up | 31.4 (17.8) | 37.9 (16.6)
  3 Month Follow-Up | 21.2 (12.6) | 32.3 (17.1)

2. Primary Outcome: Quality of Life Enjoyment and Satisfaction Questionnaire (QLESQ)
Description: The 16-item QLESQ (short form) evaluates quality of life and other areas of change related to functioning outside of symptom domains (e.g., physical health, mood, leisure time activities, social relationships, etc.). Items are rated on how satisfied the respondent has been in the past week (1 = "very poor" to 5 = "very good "). A total raw score (range: 16-80). Higher outcomes indicate better quality of life, greater enjoyment, and satisfaction.
Time Frame: Baseline, Endpoint (2 weeks after VR session 6), 1 Month Follow-Up, 3 Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 35.9 (8.9) | 39.2 (9.8)
  Endpoint | 39.2 (10.2) | 41.6 (9.2)
  1 month follow-up | 40.7 (10.3) | 41.0 (8.5)
  3-month follow-up | 44.3 (9.6) | 47.1 (10.1)

3. Primary Outcome: Psychophysiology (Skin Conductance Reactivity; SCR)
Description: Psychophysiology will include skin conductance reactivity to specific trauma context virtual reality (VR) cues presented in the VR scenario. SCR to VR events will be measured by the phasic responses that occur after the presentation of discreet VR events. SCR will be compared from baseline to end of tDCS+VR, to correlate these measures and evaluate changes attributable to active tDCS+VR compared to sham.
Time Frame: Measured during each tDCS+VR session, each session up to 1 hour
Measure: Mean (Standard Error); unit: microsiemens (μS)
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 26 | 28
microsiemens (μS)
  VR Session 1 | 0.742 (0.093) | 0.64 (0.093)
  VR Session 2 | 0.596 (0.095) | 0.503 (0.092)
  VR Session 3 | 0.48 (0.095) | 0.539 (0.093)
  VR Session 4 | 0.458 (0.096) | 0.475 (0.093)
  VR Session 5 | 0.295 (0.095) | 0.492 (0.094)
  VR Session 6 | 0.441 (0.096) | 0.492 (0.094)

4. Secondary Outcome: Inventory of Depressive Symptomatology Self-Report (IDSSR)
Description: The 28-item IDSSR is a self-report measure of depressive symptom severity. Each item is rated on a scale of 0 to 3 by the participant for a total minimum score of 0 and a maximum score of 84. A higher score on the IDSSR indicates increased depressive symptom severity.
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 41.6 (12.0) | 38.6 (13.0)
  Midpoint | 35.5 (10.7) | 35.3 (13.4)
  Endpoint | 34.2 (15.1) | 34.8 (14.5)
  1 Month Follow-Up | 30.5 (16.2) | 32.3 (15.5)
  3 Month Follow-Up | 23.4 (12.7) | 27.1 (14.8)

5. Secondary Outcome: Social and Occupational Function Scale (SOFAS)
Description: The SOFAS is a scale that focuses on the individual's level of social and occupational functioning and is not directly influenced by the overall severity of the individual's psychological symptoms. Any impairment in social and occupational functioning that is due to general medical conditions is considered in making the SOFAS rating. The SOFAS is usually used to rate functioning for the current period (i.e., the level of functioning at the time of the evaluation). Scores range from 0 to 100, with higher scores indicating better social and occupational functioning.
Time Frame: Baseline, Endpoint (2 weeks after VR session 6), 1 Month Follow-Up, 3 Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 40.5 (9.7) | 43.0 (11.2)
  Endpoint | 47.2 (14.7) | 48.0 (12.2)
  1 Month Follow-Up | 53.1 (13.8) | 54.1 (15.4)
  3 Month Follow-Up | 67.2 (8.3) | 62.2 (15.3)

6. Secondary Outcome: Clinician Administered PTSD Scale for the DSM-5 (CAPS-5)
Description: The CAPS-5 is the gold standard in clinician-assessed PTSD symptoms. The CAPS-5 is a 30-item structured interview that can be used to make current (past month) diagnosis of PTSD, make lifetime diagnosis of PTSD, and assess PTSD symptoms over the past week. In addition to assessing the 20 DSM-5 PTSD symptoms, questions target the onset and duration of symptoms, subjective distress, impact of symptoms on social and occupational functioning, improvement in symptoms since a previous CAPS administration, overall response validity, overall PTSD severity, and specifications for the dissociative subtype (depersonalization and derealization). An interviewee's total severity score on the CAPS-5 represents the sum of the individual severity scores (0-4) for each of the 20 PTSD symptoms; total scores range from 0-80, with higher scores indicating more severe PTSD symptoms.
Time Frame: Baseline, Endpoint (2 weeks after VR session 6), 1 Month Follow-Up, 3 Month Follow-Up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active Stimulation | Sham Stimulation
Number analyzed (Participants) | 26 | 28
score on a scale
  Baseline | 44.8 (8.2) | 40.5 (8.1)
  Endpoint | 40.4 (11.2) | 37.1 (9.2)
  1 Month Follow-Up | 34.1 (14.7) | 36.1 (12.6)
  3 Month Follow-Up | 22.7 (13.9) | 31 (11.9)

ADVERSE EVENTS:
Time Frame: Up to three months
Description: Adverse events were spontaneously reported by participants and systematically assessed through a side effects questionnaire that was administered before and after each tDCS + virtual reality session.
Arm/Group | Active Stimulation | Sham Stimulation
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/26 | 2/28
Other Adverse Events (participants affected / at risk) | 18/26 | 18/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Stimulation (N=26) | Sham Stimulation (N=28)
Exacerbation of chronic gastrointestinal illness (Gastrointestinal disorders) | 2 (2) | 0 (0)
Syncopal episode (General disorders) | 0 (0) | 1 (1)
Treatment-emergent suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Active Stimulation (N=26) | Sham Stimulation (N=28)
Headache (Nervous system disorders) | 5 | 11
Neck pain (General disorders) | 5 | 6
Head pain (General disorders) | 2 | 3
Scalp pain (General disorders) | 5 | 1
Tingling (General disorders) | 18 | 16
Itching (Skin and subcutaneous tissue disorders) | 17 | 7
Burning (Skin and subcutaneous tissue disorders) | 13 | 8
Redness (Skin and subcutaneous tissue disorders) | 15 | 10
Ringing or buzzing in ears (General disorders) | 4 | 8
Change in mood (Psychiatric disorders) | 11 | 18
Changes in concentration (General disorders) | 8 | 12
Sleepy, drowsy, or fatigue (General disorders) | 9 | 13
Flickering lights (General disorders) | 1 | 0
Blurry vision (General disorders) | 4 | 7
Dizziness or lightheadedness (General disorders) | 2 | 8
Nausea (General disorders) | 4 | 10

LIMITATIONS AND CAVEATS:
The COVID-19 pandemic significantly impacted recruitment, retention (particularly at the 3-month timepoint), and plausibly outcomes related to quality of life and social and occupational function.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/60/NCT03372460/Prot_SAP_000.pdf
  • Informed Consent Form (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/60/NCT03372460/ICF_001.pdf